CLINICAL TRIAL: NCT03710109
Title: Evaluation of an EEG Based Concussion System
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Putrino, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 18-0699
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Concussion
Keywords: Concussion; Sports Concussion; Sports Medicine; Electroencephalography; Steady state visual evoked potential; Evoked Potential
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Concussion: Individuals who have sustained a recent concussion
  Interventions: Other: EEG
- Control Healthy Volunteers: No Intervention

INTERVENTIONS:
Other: EEG — non-invasive, non-interventional sensor
  Groups: Concussion

SUMMARY:
This study will evaluate the accuracy of a new concussion system at detecting concussions. The investigators will be evaluating the degree to which data collected with the device agrees with a physician's determination of a concussion. The system captures an electroencephalograph (EEG) potential when a light is flashed into the eyes of an individual. The device is not FDA approved, but it is a non-significant risk device. The device is a non-invasive, non-interventional sensor. It will not replace the opinion of the physician in diagnosing a concussion.

This study will test the EEG based concussion system on 200 individuals, Participants will be made up of individuals who are seeking medical consultation at the Play Safe Concussion Clinic (10 Union Square E, New York, NY 10003) or at Mount Sinai Hospital (1468 Madison Ave, New York, NY 10029) after experiencing a head trauma. The Play Safe Clinic treats patients who reach out to Mount Sinai Physicians via the Play Safe telephone number: 212 241 2221. The doctors who see patients these locations will be involved in conducting this research. In addition to the standard-of-care clinical assessments, participants will also receive an evaluation from the concussion based system.

When a subject experiences a head trauma, the subject will be evaluated for a concussion by both the standard-of-care clinical assessments. The treating physician will provide all necessary standard-of-care evaluations and diagnostic procedures needed to properly diagnose and treat each patient and by the new concussion system. The researchers will also collect data from healthy, age-matched controls in order to collect a database of healthy responses to the technology.

To determine how accurate the new concussion system is at detecting concussions, the research team will compare the diagnostic results from the device to the diagnostic results of the doctor's assessments. The goal of this study is to develop a device that can give sound advice as to whether an individual should seek medical attention for a possible concussion following a head injury.

ELIGIBILITY:
Inclusion Criteria:

* Individuals seeking medical care Mount Sinai Hospital after sustaining a possible concussion.
* Healthy Individuals with no recent history of head trauma

Exclusion Criteria:

* Known history of epilepsy or any other seizure disorder
* Legally blind
* Reduced capacity to consent if there is not a Legally Authorized Representative (LAR) present

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals seeking medical attention at the Mount Sinai Hospital System after experiencing a head injury
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Steady State Visual Evoked Potential | up to 28 days
  the presence or absence of a steady state visual evoked potential (SSVEP)

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PT, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai Beth Israel Hospital, New York, New York
  - Abilities Research Center, New York, New York

IPD SHARING:
Plan to Share IPD: No